CLINICAL TRIAL: NCT05264909
Title: Assessment of Transcranial Electrical Stimulation and Auditory Stimulation During Walking in Parkinson Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Corporación de Rehabilitación Club de Leones Cruz del Sur (Other)
Collaborators: Colombian School of Engineering Julio Garavito (Other); Universidad del Rosario (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CorporacionRCLCS0006
Record Dates: First submitted 2022-02-22; First posted 2022-03-03 (Actual); Last update posted 2022-03-18 (Actual); Status verified 2022-02

CONDITIONS: Parkinson Disease
Keywords: transcranial direct current stimulation; auditory stimulation; gait analisys; Parkinson Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Transcranial Direct Current Stimulation TDCS (Experimental): Each subject will receive transcranial electrical stimulation at primary motor located in Cz based on the EEG 10-20 international system. The program include 18 sessions with a frequency of 3 times per week during 6 weeks. Therefore, during tDCS sessions, subjects will receive stimulation for 15 minutes with a current of 1.5 milliamp using 7x5 cm electrodes.
  During the stimulation, the patient must simultaneously perform gait training for 30 minutes where the speed of each step is guided by the frequency of biaural rhythms and beats, constantly heard through hearing aids. Additionally, the length of the passage will be indicated by white stripes (50 cm long and 5 cm wide), placed perpendicular along a walkway of 6.5 m.
  Thus, each session will be monitored on safety aspects of the subjects with emphasis on skin problems and other possible side effects of tDCS.
  Interventions: Device: Multi-channel Transcranial direct current stimulation

INTERVENTIONS:
Device: Multi-channel Transcranial direct current stimulation — A medical grade tDCS device will be use in this study (Star Stim TES, Neuroelectrics, Spain). The device is a wireless multi-channel transcranial direct current stimulator that incorporates an 8-channel headcap for stimulation through gel electrodes or classic sponge electrodes. The device is integrated with a user interface for the configuration and monitoring of the stimulus parameters and a fast multifocal simulation of the tDCS electric field using an advanced brain model

SUMMARY:
Parkinson's disease affects 1 in 100 people over the age of 60. Parkinson's disease (PD) is a progressive disease of the nervous system that affects movement, produced by the destruction of dopaminergic neurons found in a region of the brain called the basal ganglia Over time, different strategies have been developed to treat and slow the progress of the disease, including pharmacological, rehabilitative and even surgical treatments.

Transcranial direct current stimulation (tDCS) is a brain stimulation technique that delivers a low-intensity electrical current to the scalp, usually between 1 and 2 mA over approximately 5 to 30 minutes. The tDCS technique is used with the aim of enhancing a specific brain activity through the neuromodulation of neuronal excitability. In pathologies such as PD, these therapies have been shown to induce immediate after-effects in the brain that translate into reduced gait freezing and improvements in executive function and mobility. In addition, the combined effects of tDCS and physical therapy on the walking ability of PD patients have been studied, where it was shown that anodic tDCS and physiotherapy could be used as a combination treatment to improve patients' gait speed.

Another potential therapeutic tool in the treatment of PD consists of the use of sound stimulation with beat frequencies similar to the step. Specifically, this technology is characterized by presenting two tones of different frequencies for each ear in order to influence the mood and mental performance of the listener.

This protocol is proposed in order to evaluate the effect of tDCS combined with auditory and binaural stimulus strategies during gait therapy in patients with Parkinson's disease.

DETAILED DESCRIPTION:
According to the World Health Organization (WHO), Parkinson's disease affects 1 in 100 people over the age of 60. Currently, there are about 7 million people with this disease in the world and the WHO predicts that by 2030 they will reach more than 12 million.

Parkinson's disease (PD) is a progressive disease of the nervous system that affects movement, produced by the destruction of dopaminergic neurons found in a region of the brain called the basal ganglia. This disease usually affects people over 60 years of age, whose symptoms worsen as the disease progresses and in many cases the ability to function in everyday situations is greatly affected. Due to decreased levels of dopamine, motor symptoms such as tremor, stiffness, slowness of movement, postural instability and other non-motor symptoms such as depression, hallucinations, insomnia and dysfunction of the autonomous organic systems, for example, digestion and blood pressure, as well as alteration in the expression of emotions. Over time, different strategies have been developed to treat and slow the progress of the disease, including pharmacological, rehabilitative and even surgical treatments.

Transcranial direct current stimulation (tDCS) is a brain stimulation technique that delivers a low-intensity electrical current to the scalp, usually between 1 and 2 mA over approximately 5 to 30 minutes. During tDCS, most people feel a slight tingling, pricking, itching or warmth, however, these sensations are not painful and disappear when the stimulation is stopped. The tDCS technique is used with the aim of enhancing a specific brain activity through the neuromodulation of neuronal excitability. In pathologies such as PD, these therapies have been shown to induce immediate after-effects in the brain that translate into reduced gait freezing and improvements in executive function and mobility. In addition, the combined effects of tDCS and physical therapy on the walking ability of PD patients have been studied, where it was shown that anodic tDCS and physiotherapy could be used as a combination treatment to improve patients' gait speed.

Another potential therapeutic tool in the treatment of PD consists of the use of sound stimulation with beat frequencies similar to the step. Sounds, mainly rhythm, have also been shown to improve gait characteristics (speed, time and cadence of passage) and eliminate frozen gait, characteristic in this type of population. Sound strategies such as Binaural Beats (BBs) improve the ability of upper and lower limb movements in PD patients. Specifically, this technology is characterized by presenting two tones of different frequencies for each ear in order to influence the mood and mental performance of the listener. In accordance with the above, this protocol is proposed in order to evaluate the effect of tDCS combined with auditory and binaural stimulus strategies during gait therapy in patients with Parkinson's disease.

ELIGIBILITY:
Inclusion Criteria:

* Parkinson Disease
* Both gender
* Informed consent accepted
* Adults

Exclusion Criteria:

* Mental diseases
* Injuries in the scalp skin
* Inflammatory tegumentary diseases
* Migraines
* Pregnancy

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Estimated)
Dates: Start 2021-08-01 (Actual); Primary Completion 2022-12-01 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Gait Deviation Index Baseline | Baseline
  Gait Deviation Index will be calculated for each patient using a 3D VICON infra-red camera system
Gait Deviation Index Post-Intervention | 8 weeks
  Gait Deviation Index will be calculated for each patient using a 3D VICON infra-red camera system

SECONDARY OUTCOMES:
Power spectral density in the frequency of motor imagery from primary motor cortex Baseline | Baseline
  continuous signals will be acquired from the primary motor cortex of lower limbs (FcZ, C2, Cz, C1, Cpz) according to the 10-20 International EEG System. Power spectral density in the frequency band of motor imagery (8-32Hz) will be obtained by OpenVibe Software and Matlab. The measure unit is Decibels per Hertz(dB/Hz).
Power spectral density in the frequency of motor imagery from primary motor cortex Post-Intervention | 8 weeks
  continuous signals will be acquired from the primary motor cortex of lower limbs (FcZ, C2, Cz, C1, Cpz) according to the 10-20 International EEG System. Power spectral density in the frequency band of motor imagery (8-32Hz) will be obtained by OpenVibe Software and Matlab. The measure unit is Decibels per Hertz(dB/Hz).

CONTACTS AND LOCATIONS:
Overall Officials: Patricio E Barría Aburto, MSc., Principal Investigator — Corporación de Rehabilitacion Club de Leones Cruz del Sur
Locations (1):
- Corporación de Rehabilitación Club de Leones Cruz del Sur, Punta Arenas, Region of Magallanes, Chile

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Areas FZDS, Nakamura-Palacios EM, Boening A, Areas GPT, Nascimento LR. Does neuromodulation transcranial direct current stimulation (tDCS) associated with peripheral stimulation through exercise to walk have an impact on falls in people with Parkinson's disease? Med Hypotheses. 2020 Nov;144:109916. doi: 10.1016/j.mehy.2020.109916. Epub 2020 Jun 4. PMID 32526508
- [Background] Dagan M, Herman T, Harrison R, Zhou J, Giladi N, Ruffini G, Manor B, Hausdorff JM. Multitarget transcranial direct current stimulation for freezing of gait in Parkinson's disease. Mov Disord. 2018 Apr;33(4):642-646. doi: 10.1002/mds.27300. Epub 2018 Feb 13. PMID 29436740
- [Background] Yotnuengnit P, Bhidayasiri R, Donkhan R, Chaluaysrimuang J, Piravej K. Effects of Transcranial Direct Current Stimulation Plus Physical Therapy on Gait in Patients With Parkinson Disease: A Randomized Controlled Trial. Am J Phys Med Rehabil. 2018 Jan;97(1):7-15. doi: 10.1097/PHM.0000000000000783. PMID 28650857
- [Background] Ghai S, Ghai I, Schmitz G, Effenberg AO. Effect of rhythmic auditory cueing on parkinsonian gait: A systematic review and meta-analysis. Sci Rep. 2018 Jan 11;8(1):506. doi: 10.1038/s41598-017-16232-5. PMID 29323122
- [Background] Brabenec L, Klobusiakova P, Barton M, Mekyska J, Galaz Z, Zvoncak V, Kiska T, Mucha J, Smekal Z, Kostalova M, Rektorova I. Non-invasive stimulation of the auditory feedback area for improved articulation in Parkinson's disease. Parkinsonism Relat Disord. 2019 Apr;61:187-192. doi: 10.1016/j.parkreldis.2018.10.011. Epub 2018 Oct 10. PMID 30337204
- [Background] Galvez G, Recuero M, Canuet L, Del-Pozo F. Short-Term Effects of Binaural Beats on EEG Power, Functional Connectivity, Cognition, Gait and Anxiety in Parkinson's Disease. Int J Neural Syst. 2018 Jun;28(5):1750055. doi: 10.1142/S0129065717500551. Epub 2017 Nov 13. PMID 29297265
- [Background] Costa-Ribeiro A, Maux A, Bosford T, Aoki Y, Castro R, Baltar A, Shirahige L, Moura Filho A, Nitsche MA, Monte-Silva K. Transcranial direct current stimulation associated with gait training in Parkinson's disease: A pilot randomized clinical trial. Dev Neurorehabil. 2017 Apr;20(3):121-128. doi: 10.3109/17518423.2015.1131755. Epub 2016 Feb 10. PMID 26864140
- [Background] Galli M, Cimolin V, De Pandis MF, Schwartz MH, Albertini G. Use of the Gait Deviation index for the evaluation of patients with Parkinson's disease. J Mot Behav. 2012;44(3):161-7. doi: 10.1080/00222895.2012.664180. Epub 2012 Mar 28. PMID 22455905
- [Background] Stuart S, Wagner J, Makeig S, Mancini M. Brain Activity Response to Visual Cues for Gait Impairment in Parkinson's Disease: An EEG Study. Neurorehabil Neural Repair. 2021 Nov;35(11):996-1009. doi: 10.1177/15459683211041317. Epub 2021 Sep 10. PMID 34505536